

#### STATISTICAL ANALYSIS PLAN

**Study Title:** A Phase 2, Open-label Study to Investigate the Efficacy and

Safety of Ledipasvir/Sofosbuvir Fixed Dose Combination in the Treatment of Hepatitis C Virus (HCV) Infection in Pediatric Subjects Undergoing Cancer Chemotherapy

Name of Test Drug: Ledipasvir/Sofosbuvir Fixed-Dose Combination

(LDV/SOF FDC)

Study Number: GS-US-337-1904

**Protocol Version (Date):** Original: 06 Oct 2015

Amendment 1.0: 16 June 2017

**Analysis Type:** Final Analyses

**Analysis Plan Version:** 1.0

**Analysis Plan Date:** 01 Mar 2019

Analysis Plan Author: PPD

#### CONFIDENTIAL AND PROPRIETARY INFORMATION

## TABLE OF CONTENTS

| TAI | BLE O | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF A | ABBREVIATIONS | 4 |
| 1. | INTR | RODUCTION | 6 |
| | 1.1.<br>1.2.<br>1.3. | Study Objectives Study Design Sample Size and Power | 7 |
| 2. | TYPE | E OF PLANNED ANALYSIS | 8 |
| | 2.1.<br>2.2.<br>2.3. | Data Monitoring Committee Interim Analysis Final Analysis | 8<br>8 |
| 3. | GENI | ERAL CONSIDERATIONS FOR DATA ANALYSES | 9 |
| | 3.1. | Analysis Sets 3.1.1. All Enrolled Analysis Set 3.1.2. Full Analysis Set 3.1.3. Safety Analysis Set | 9<br>9 |
| | 3.2.<br>3.3.<br>3.4.<br>3.5. | Subject Grouping | 9<br>9 |
| | 3.6. | 3.5.1. Missing Data 3.5.2. Outliers | 10<br>11 |
| | 3.7. | Visit Windows 3.7.1. Definition of Study Day 3.7.2. Analysis Windows 3.7.3. Selection of Data in the Event of Multiple Records in an Analysis Window | 12<br>12<br>13 |
| 4. | SUBJ | JECT DISPOSITION | 15 |
| | 4.1.<br>4.2. | Subject Enrollment and Disposition Extent of Exposure 4.2.1. Duration of Exposure to Study Drug 4.2.2. Adherence to Study Drug | 16<br>16 |
| | 4.3. | Protocol Deviations | |
| 5. | | | 18 |
| | 5.1.<br>5.2.<br>5.3.<br>5.4. | Demographics Other Baseline Characteristics Swallowability Assessment for LDV/SOF Tablets Medical History | 18<br>19 |
| 6. | EFFICACY ANALYSES | | |
| | 6.1. | Primary Efficacy Endpoint | 20<br>20 |
| | 6.2. | Secondary Efficacy Endpoints 6.2.1. Definition of Secondary Efficacy Endpoints 6.2.2. Analysis Methods for Secondary Efficacy Endpoints | 20<br>20 |
| | 6.3 | Exploratory Endpoints of Interest | 22 |

| | | 6.3.1. | Definition of Exploratory Endpoints | 22 |
|---|---|---|---|---|
| | | 6.3.2. | Analysis Methods for Other Endpoints of Interest | 22 |
| | 6.4. | Changes | s From Protocol-Specified Efficacy Analyses | 23 |
| 7. | SAFE | ΓΥ ANAI | LYSES | 24 |
| | 7.1. | Adverse | Events and Deaths | 24 |
| | | 7.1.1. | Adverse Event Dictionary | |
| | | 7.1.2. | Adverse Event Severity | |
| | | 7.1.3. | Relationship of Adverse Events to Study Drug | |
| | | 7.1.4. | Serious Adverse Events | |
| | | 7.1.5. | Treatment-Emergent Adverse Events | |
| | | | 7.1.5.1. Definition of Treatment Emergent | |
| | | <b>5</b> 16 | 7.1.5.2. Incomplete Dates | |
| | 7.0 | 7.1.6. | Summaries of Adverse Events and Deaths | |
| | 7.2. | | ory Evaluations | |
| | | 7.2.1.<br>7.2.2. | APRI Calculation | |
| | | 7.2.2. | Graded Laboratory Values | |
| | | 1.2.3. | 7.2.3.1. Treatment-Emergent Laboratory Abnormalities | |
| | | | 7.2.3.2. Summaries of Laboratory Abnormalities | |
| | 7.3. | Body W | eight, Height, and Vital Signs | |
| | 7.4. | d Concomitant Medications. | | |
| | | 7.4.1. | Prior Medications | |
| | | 7.4.2. | Concomitant Medications | 29 |
| | 7.5. | | afety Measures | |
| | 7.6. | Changes | s From Protocol-Specified Safety Analyses | 30 |
| 8. | PHAR | MACOK | INETIC ANALYSES | 31 |
| 9. | REFEI | RENCES | | 32 |
| 10. | SOFT | WARE | | 33 |
| 11. | | | 1 | |
| 12. | APPENDICES | | | |
| 12. | ALL | NDICES. | | |
| | Appen | ıdix 1. | Schedule of Assessments | 36 |
| | | | LIST OF IN-TEXT-TABLES | |
| | Table : | Analysis Windows for On-treatment HCV RNA, Vital Signs, Height and | | |
| | | | Weight, Fibrotest a, and Safety Laboratory Data | 13 |
| | Table : | 3-2. | Analysis Windows for Posttreatment HCV RNA, Vital Sign, Height and | |
| | | | Weight, FibroScan, Fibrotest, and Safety Laboratory Data | 13 |

#### LIST OF ABBREVIATIONS

٠

AE adverse event

ALT alanine aminotransferase
APRI AST to Platelet Ratio Index

APTT activated partial thromboplastin time

AST aspartate aminotransferase BLQ below the limit of quantitation

BMI body mass index

CFR Code of Federal Regulations

CI confidence interval
CrCL Creatinine clearance
CRF case report form
CSR clinical study report

dL deciliter

DMC data monitoring committee

EC Ethnic Committee
ECG electrocardiogram

eCRF electronic case report form(s)

EOT End of Treatment

ESDD Early Study Drug Discontinuation

FAS full analysis set

FDC fixed-dose combination

FU follow-up

Gilead Gilead Sciences, Inc.

HCV hepatitis C virus

HLGT high-level group term

HLT high level term

ICH International Conference on Harmonization (of Technical Requirements for Registration of

Pharmaceuticals for Human Use)

ID identification

INR International Normalized Ratio of prothrombin time

LDV ledipasvir

LDV/SOF ledipasvir/sofosbuvir LLT lower level term

LLOQ lower limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

NCI National Cancer Institute, Egypt

PK pharmacokinetics
PT preferred term
Q1 first quartile

| third quartile |
|----------------------------------------------------------------|
| red blood cell |
| ribonucleic acid |
| serious adverse event |
| statistical analysis plan |
| statistical analysis software |
| standard deviation |
| standard error |
| International system of units |
| system organ class |
| sofosbuvir |
| sustained virologic response |
| sustained virologic response x weeks after stopping study drug |
| Treatment-emergent adverse events |
| tables, figures, and listings |
| target not detected |
| upper limit of normal |
| white blood cell |
| World Health Organization |

## 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the clinical study report (CSR) for Study GS-US-337-1904. This SAP is based on the protocol amendment 1.0 16 June 2017. Related documents are the original study protocol and electronic case report form (eCRF). The SAP will be finalized before database finalization. Any changes made after the finalization of the SAP will be documented in the CSR.

An interim analysis for safety was performed after a total of 11 subjects had completed Week 12 assessment or prematurely discontinued from the study before proceeding to recruitment of remaining subjects. The purpose of this interim analysis was to respond to EC committee request of safety concern on pediatric population.

## 1.1. Study Objectives

The primary objective of this study is as follows:

- To evaluate the efficacy of ledipasvir/sofosbuvir (LDV/SOF) in treating HCV infection in pediatric subjects who are undergoing cancer chemotherapy, as measured by the proportion who achieve a sustained virologic response 12 weeks after the end of HCV treatment (SVR12)
- To evaluate the safety and tolerability of treatment with LDV/SOF for 12 weeks

The secondary objectives of this study are as follows:

- To determine the proportion of subjects who attain SVR at 4 and 24 weeks after cessation of HCV treatment (SVR4 and SVR24)
- To evaluate the kinetics of circulating HCV RNA during treatment and after cessation of HCV treatment

The exploratory objectives of this study are:





This is a phase 2 single-center open-label study investigating the efficacy and safety of LDV/SOF FDC in pediatric subjects with chronic HCV who are receiving maintenance cancer chemotherapy.

Approximately 40 treatment naïve or experienced pediatric subjects will be enrolled in this study. Male and female children 12 to < 18 years of age, with genotype 1 or 4 HCV infection, and who are receiving a maintenance cancer chemotherapy regimen will be enrolled.

All subjects will receive LDV/SOF FDC once daily with or without food for 12 weeks. Subjects will be assigned to receive 1 LDV/SOF FDC 90 mg/ 400 mg tablet daily or 4 LDV/SOF FDC 22.5 mg/100 mg tablets once daily based on a swallowability assessment performed at screening up to Day 1.

Subjects who have indicated that they can take pills will be observed taking a placebo to match the 90 mg/ 400 mg LDV/SOF FDC tablet. If a subject is unable to swallow the 90 mg/ 400 mg LDV/SOF FDC tablet size, he/she will repeat the assessment with a placebo to match the 22.5 mg/ 100 mg LDV/SOF FDC tablet. If unable to swallow the 22.5 mg/ 100 mg LDV/SOF FDC tablet, the subject will be screen failed and excluded from the study.

The total time to complete all study visits is up to approximately 40 weeks including the following periods:

- 28-day (4-week) screening period
- 12-week treatment period
- Up to 24-week posttreatment period

The schedule of assessments is provided as an appendix to the SAP (**Appendix 1**).

#### 1.3. Sample Size and Power

With approximately 40 subjects enrolled into the study, a 2-sided 95% confidence interval of the SVR12 rate will extend at most 26.6% in length, assuming the expected SVR12 rate is 80%.

The study was terminated after 19 subjects were enrolled due to extremely slow enrollment rate.

#### 2. TYPE OF PLANNED ANALYSIS

## **2.1.** Data Monitoring Committee

This study does not have a data monitoring committee (DMC).

## 2.2. Interim Analysis

There was 1 planned interim safety analysis after 11 subjects had completed Week 12 assessment or prematurely discontinued from the study before proceeding to recruitment of remaining subjects. Decision to continue recruitment of remaining subjects was contingent on review of safety data (adverse events and laboratory abnormalities) from the first 11 subjects who completed the treatment period.

No formal interim efficacy analysis with the possibility of early termination for efficacy or futility is planned.

## 2.3. Final Analysis

The final analysis will be conducted when all subjects have completed the 24 week post treatment visit or prematurely discontinued from the study. The data will be finalized after all data queries are resolved for study visits through completion of the 24-week posttreatment visit. At the conclusion of data finalization, the study statistician and statistical programmers will run the final version TFLs.

## 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects [n], mean, standard deviation [SD] or standard error [SE], median, first quartile [Q1], third quartile [Q3], minimum, and maximum will be presented.

Data collected in the study will be presented in by-subject listings for all subjects in the Safety Analysis Set, unless otherwise specified. All by-subject listings will be presented by subject identification (ID) number in ascending order, unless otherwise specified.

## 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. The number of subjects eligible for each analysis set will be provided. Subjects who were excluded from each analysis set will be summarized or provided in a by-subject listing with reasons for exclusion.

### 3.1.1. All Enrolled Analysis Set

All Enrolled Analysis Set includes all subjects enrolled in the study after screening.

### 3.1.2. Full Analysis Set

The Full Analysis Set (FAS) includes all enrolled subjects who took at least 1 dose of study drug. The study drug in this study is LDV/SOF FDC.

This is the primary analysis set for efficacy analyses.

#### 3.1.3. Safety Analysis Set

The Safety Analysis Set includes all subjects who took at least 1 dose of study drug. This is the primary analysis set for safety analyses.

#### 3.2. Subject Grouping

This is a single arm study. All subjects received LDV/SOF 90mg/400mg daily for 12 weeks (including 90/400mg tablet or 4 22.5/100mg tablets).

#### 3.3. Strata and Covariates

This study does not use a stratified randomization schedule for enrolling subjects.

#### 3.4. Examination of Subject Subsets

The primary efficacy endpoint, SVR12, will be analyzed for the following subsets:

• Age group ( $\geq 12$ -  $\leq 15$  years old,  $\geq 15$  years old)

- Sex (male, female)
- baseline weight (<= median, > median)
- IL28B (CC, non-CC; with non-CC further broken down to CT, TT)
- cirrhosis (presence, absence, missing)
- HCV genotype subtypes (4a, 4b, 4c or 4d, 4h etc.)
- baseline HCV RNA (< 800,000, ≥800,000 IU/mL)
- baseline alanine aminotransferase (ALT) ( $\leq 1.5 \times \text{upper limit of normal (ULN)}$ ,  $> 1.5 \times \text{ULN}$ )
- prior HCV treatment (treatment naive, treatment experienced)
- most recent HCV treatment response (non-responder, relapse/breakthrough, Other) for treatment-experienced subjects
- study treatment status (completed study treatment, discontinued study treatment)
- adherence to study regimen (<80%,  $\ge80\%$ )

## 3.5. Missing Data and Outliers

#### 3.5.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified.

For missing last dose date of study drug, imputation rules are described in Section 3.7.1. The handling of missing or incomplete dates for AE onset is described in Section 7.1.5.2, and for prior and concomitant medications in Section 7.4.

For analyses of categorical HCV RNA data, missing posttreatment HCV RNA data will have the missing data imputed. Missing on-treatment HCV RNA will have the missing data imputed up to the time of the last dose (for on-treatment displays). If the study day associated with the last dosing date is greater than or equal to the lower bound of a visit window, and the value at the visit is missing, the value will be imputed. If the study day associated with the last dosing date is less than the lower bound of a visit window then the on-treatment value at that visit will remain missing.

If a data point is missing and is preceded and followed in time by values that are "< LLOQ target not detected (TND)", then the missing data point will be set to "< LLOQ TND". If a data point is missing and preceded and followed by values that are "< LLOQ detected", or proceeded by "< LLOQ detected" and followed by "< LLOQ TND", or preceded by "< LLOQ TND" and followed by "< LLOQ detected", then the missing value will be set to "<

LLOQ detected". In these situations the data point will be termed a bracketed success; otherwise, the data point will be termed a bracketed failure (ie, ≥ LLOQ detected). If a data point is missing and is not bracketed, the missing data point will also be termed a failure (ie, ≥ LLOQ detected) except for SVR24, which will be imputed according to SVR12 status. Success for SVR12 who have no further HCV RNA measurements collected will be counted as a success for SVR24 due to the high correlation between these 2 endpoints.

For the analyses of continuous HCV RNA efficacy data, when and only when a missing HCV RNA value is imputed as < LLOQ TND or < LLOQ detected according to the imputation rule described above, the corresponding continuous value will be imputed to LLOQ - 1 IU/mL. No other imputation will be performed for continuous HCV RNA data.

#### 3.5.2. Outliers

Outliers will be identified during the data management and data analysis process, but no sensitivity analyses will be conducted. All data will be included in the data analysis.

### 3.6. Data Handling Conventions and Transformations

By-subject listings will be presented for all subjects in the Safety Analysis Set sorted by subject ID number, visit date, and time (if applicable) unless otherwise specified. Data collected on log forms, such as AEs, will be presented in chronological order within subject.

Age (in years) on the date of the first dose of study drug will be used for analyses and presentation in listings.

If a subject was not dosed with study drug at all, then the date the informed consent was signed will be used instead of the first dose date of study drug.

Data that are continuous in nature but are less than the lower limit of quantitation or above the upper limit of quantitation will be imputed as follows:

- A value that is one unit less than the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "< x" (where x is considered the limit of quantitation). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used for calculation of summary statistics. An exception for this rule is any value reported < 1. For the values reported as < 1 or < 0.1, value of 0.9 or 0.09 will be used for calculation of summary statistics.
- A value that is one unit above the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "> x" (where x is considered the limit of quantitation). Values with decimal points will follow the same logic as above.
- The limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the limit of quantitation).

The artus® HCV RG RT-PCR Kit by QIAGEN March 2015 was used to determine HCV RNA results in this study. The lower limit of quantitation (LLOQ) of this assay is 50 IU/mL.

When the calculated IU/mL is within the linear range of the assay, then the result will be reported as the "<< numeric value>> IU/mL". This result will be referred to in this document as the numeric result or as "> LLOO detected" for categorical result.

When HCV RNA is not detected, the result is reported as "HCV RNA not detected" or "target not detected". This result will be referred to in this document as "< LLOQ target not detected" or "< LLOQ TND".

When the HCV RNA IU/mL is less than LLOQ of the assay, the result is reported as "<50 IU/mL HCV RNA detected". This result will be referred to in this document as "< LLOQ detected".

The overall category of HCV RNA < LLOQ includes "< LLOQ TND" and "< LLOQ detected."

For numerical HCV RNA data, values below LLOQ will be set to the LLOQ – 1 IU/mL. (ie, 49 HCV RNA IU/mL). HCV RNA values returned as "No HCV RNA detected" will also be set to 49 IU/mL.

For selected analyses, HCV RNA data (IU/mL) will be transformed to the logarithmic (base 10) scale (log<sub>10</sub> IU/mL).

#### 3.7. Visit Windows

#### 3.7.1. Definition of Study Day

Study day is the day relative to the date of the first dose of study drug. Study Day 1 will be defined as the day of first dose of study drug administration.

Study day will be calculated from the date of first dose of study drug administration and derived as follows:

- For postdose study days: Assessment Date First Dose Date + 1
- For days prior to the first dose: Assessment Date First Dose Date

The last dose date for an individual study drug will be the end date on study drug administration eCRF for the record where the "subject permanently discontinued" flag is 'Yes'. The last dose date will be defined as the maximum of the last dose dates of individual study drugs in a treatment group.

If there are subjects for whom the date of last study drug is unknown due to the reason that the subject was lost to follow-up and not able to be contacted, the date of last dose will be estimated using the maximum of nonmissing study drug start or stop dates, visit dates and laboratory collection dates (posttreatment visits and unscheduled visits are not included).

## 3.7.2. Analysis Windows

Subject visits might not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows. In general, the baseline value will be the last nonmissing value on or prior to the first dose date of study drug.

Safety laboratory data, HCV RNA, vital signs, height and weight, FibroScan, and Fibrotest, collected up to the last dose date + 3 days are considered to be on-treatment data. The analysis windows for on-treatment HCV RNA, vital signs, height and weight, and safety laboratory data are provided in Table 3-1.

Table 3-1. Analysis Windows for On-treatment HCV RNA, Vital Signs, Height and Weight, Fibrotest <sup>a</sup>, and Safety Laboratory Data

| Nominal Visit | Nominal Day | Lower Limit | Upper Limit |
|---------------|-------------|-------------|-------------|
| Baseline | 1 | (none) | 1 |
| Week 1 | 7 | 2 | 11 |
| Week 4 | 28 | 12 | 42 |
| Week 8 | 56 | 43 | 70 |
| Week 12 | 84 | 71 | ≥85 |

<sup>&</sup>lt;sup>a</sup> Analysis windows for coagulation parameters and Fibrotest are only defined for Baseline and Week 12.

Safety laboratory data, HCV RNA, vital signs, height and weight, FibroScan, and Fibrotest, collected after the last dose date + 3 days will be assigned to the posttreatment follow-up (FU) visits. Visit windows will be calculated from the last dose date (ie, FU Day = collection date minus the last dose date) as shown in Table 3-2.

Table 3-2. Analysis Windows for Posttreatment HCV RNA, Vital Sign, Height and Weight, FibroScan, Fibrotest, and Safety Laboratory Data

| | HCV RNA, He | ight and Weigh<br>and Fibrotest | t, FibroScan | Vital Signs and Safety Laboratory Data b | | |
|---|---|---|---|---|---|---|
| Nominal<br>FU <sup>a</sup> Visit | Nominal FU<br>Day | Lower<br>Limit | Upper Limit | Nominal FU<br>Day | Lower<br>Limit | Upper Limit |
| FU-4° | 28 | 21 | 69 | 28 | 4 | 30 |
| FU-12 | 84 | 70 | 146 | NA | NA | NA |
| FU-24 | 168 | 147 | 210 | NA | NA | NA |

FU-x visit = posttreatment Week-x follow-up visit.

b FibroScan is collected at screening, posttreatment week 12 and posttreatment week 24.

b Vital signs and safety labs will only be summarized for the FU-4 visit (up to 30 days after last dose).

c Doesn't apply to FibroScan and Fibrotest.

# 3.7.3. Selection of Data in the Event of Multiple Records in an Analysis Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window.

If multiple valid nonmissing numeric observations exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- For baseline, the last available record on or prior to the date of the first dose of study drug will be selected.
- For postbaseline visits:
  - The record closest to the nominal day for that visit will be selected except for HCV RNA posttreatment follow-up visits, for which the latest record in the analysis window will be selected.
  - If there are 2 records that are equidistant from the nominal day, the later record will be selected.
  - If there is more than 1 record on the selected day, the average will be taken, unless otherwise specified.
- If multiple valid nonmissing categorical observations exist in a window, records will be selected as follows:
  - For baseline, the last available record on or prior to the date of the first dose of study drug will be selected. If there are multiple records with the same time or no time recorded on the same day, the value with the lowest severity will be selected (eg, normal will be selected over abnormal).
  - For postbaseline visits, follow the same rules described above for postbaseline numeric observations, except that if there are multiple records on the same day, the most conservative value will be selected (eg, abnormal will be selected over normal).

### 4. SUBJECT DISPOSITION

## 4.1. Subject Enrollment and Disposition

A summary of subject disposition will be provided. This summary will present the number of subjects screened, the number of subjects enrolled, and the number and percentage of subjects in each of the categories listed below. For the "Treated" category, the denominator for the percentage calculation will be the total number of subjects enrolled for each column. For all other categories, the denominator for the percentage calculation will be the total number of subjects in the Safety Analysis Set for each column.

- Treated (Safety Analysis Set)
- In FAS
- Completed study treatment
- Did not complete study treatment with reason for premature discontinuation of study treatment
- Completed the study (completed posttreatment Week 24 visit)
- Did not complete the study with reason for premature discontinuation of study

Among subjects who completed study treatment and who discontinued study treatment, the number and percentage of subjects will be summarized for:

- Who had no HCV posttreatment Week 4 assessment and thereafter (No HCV FU-4 and thereafter)
- Who had HCV posttreatment Week 4 assessment but no HCV posttreatment Week 12 assessment and thereafter (With HCV FU-4 but No FU-12 and thereafter)

If a subject did not have any HCV RNA assessment  $\geq$  21 days after the last dose of any study drug (ie, lower bound of FU-4 visit for HCV RNA data), the subject is categorized as having "No HCV FU-4 and thereafter". If a subject had the HCV FU-4 assessment but did not have any HCV RNA assessment  $\geq$  70 days after the last dose of any study drug (ie, lower bound of FU-12 visit for HCV RNA data), the subject is categorized as having "With HCV FU-4 but No FU-12 and thereafter".

In addition, the total number of subjects who were enrolled in the study, and the number and percentage of subjects in each of the disposition categories listed above will be displayed in a flowchart.

The following by-subject listings will be provided by subject ID number in ascending order to support the above summary tables:

- Disposition for subjects who complete study treatment and study
- Disposition for subjects who did not complete study treatment and/or study with reasons for premature discontinuation of study drug and/or study
- Lot number and kit ID

## 4.2. Extent of Exposure

Extent of exposure to study drug will be examined by assessing the total duration of study drug exposure and the level of adherence to the study drug regimen specified in the protocol.

## **4.2.1.** Duration of Exposure to Study Drug

Total duration of exposure to study drug will be defined as last dose date minus first dose date plus 1, regardless of any temporary interruptions in study drug administration, and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks). If subjects are continuing on study drug, use the last study drug end date, clinical visit date, or laboratory visit date, whichever occurred last during the on-treatment period [or use the data cutoff date for analysis] to impute the last dose date for the calculation of the duration of study drug exposure.

The total duration of exposure to study drug will be summarized using descriptive statistics (number of subjects [n], mean, standard deviation [SD], median, first quartile [Q1], third quartile [Q3], minimum, and maximum) and using the number (ie, cumulative counts) and percentage of subjects exposed through the following time periods: Baseline (Day 1), Week 1 (Day 7); Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84). A 3-day window is applied to the last planned on-treatment visit to match with the protocol-specified visit window. Summaries will be provided for the Safety Analysis Set.

#### 4.2.2. Adherence to Study Drug

The total number of tablets administered will be summarized using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum).

The presumed total number of tablets administered to a subject will be determined by the data collected on the drug accountability CRF using the following formula:

```
Total Number of Doses Administered = (\sum No. \text{ of Tablets Dispensed}) - (\sum No. \text{ of Tablets not administered})
```

The level of adherence to the study drug regimen will be assessed based on the total amount of study drug administered relative to the total amount of study drug prescribed at baseline.

The level of adherence will be expressed in percentage using the following formula:

Level of Adherence (%) = 
$$\left(\frac{\text{Total Amount of Study Drug Administered}}{\text{Total Amount of Study Drug Prescribed at baseline}}\right) \times 100$$

Note: If calculated adherence is greater than 100%, the result will be set to 100%.

In this study, the total amount of LDV/SOF (90 mg/400 mg) prescribed for 12 weeks of treatment would require 84 tablets. For LDV/SOF (22.5 mg/ 100 mg), the total amount of tablets would be 336.

Subjects who prematurely discontinue study drug for lack of efficacy (ie, virologic failure) will have the total amount of study drug prescribed calculated up to the first date when virologic failure criteria were met. For virologic failure confirmed by 2 consecutive measurements the date of the first measurement will be used. If there are study drug bottles dispensed on or after the subject first met virologic failure criteria, these bottles will not be included in the calculation of adherence. If a bottle is dispensed and the bottle is returned empty, then the number of tablets returned will be entered as zero. If a bottle is dispensed but not returned (missing), the number of tablets taken from that bottle will be counted as zero.

Descriptive statistics for the level of adherence (n, mean, SD, median, Q1, Q3, minimum, and maximum) with the number and percentage of subjects belonging to adherence categories (eg, < 80%,  $\ge 80$  to < 90%,  $\ge 90\%$ ) will be provided for the Safety Analysis Set. No inferential statistics will be provided.

A separate by-subject listing of study drug administration and drug accountability will be provided by subject ID number (in ascending order) and visit (in chronological order).

#### 4.3. Protocol Deviations

A summary of important protocol deviations will be provided by the Clinical Operations group for subjects in the Safety Analysis Set.

## 5. BASELINE CHARACTERISTICS

## 5.1. Demographics

Subject demographic variables (ie, age, sex, race, and ethnicity) will be summarized using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) for age, and using the numbers and percentages of subjects for age categories (<= 15 years old, > 15 years old), sex, race, and ethnicity. Age is calculated in years at the date of initial study drug administration. If a subject did not receive study drug after enrollment, the subject's age will be calculated from the date that the subject signed the informed consent form. The summary of demographic data will be provided for the Safety Analysis Set.

A by-subject demographic listing will be provided by subject ID number in ascending order.

#### **5.2.** Other Baseline Characteristics

Other baseline characteristics include:

- weight in kg
- height in cm
- body mass index (BMI; in kg/m<sup>2</sup>) as a continuous variable
- IL28B (CC, Non-CC (CT, TT)
- HCV genotype and subtypes
- cirrhosis (presence, absence, unknown)
- baseline HCV RNA (log10 IU/mL) as a continuous variable and as categories < 800,000 IU/mL, ≥ 800,000 IU/mL)</li>
- baseline ALT (U/L) as a continuous variable and as categories (≤1.5 x ULN, > 1.5 x ULN)
- prior HCV treatment experience (treatment naïve or treatment experienced)
- most recent HCV treatment response (Non-Responder, Relapse/Breakthrough, other including early treatment discontinuation, met a virologic stopping rule, or unknown) for treatment-experienced subjects
- Creatinine clearance (CrCL) using the Schwartz formula as follows:

Creatinine clearance (mL/min/1.73 $m^2$ ) = k \* height (cm) / serum creatinine (mg/dL) where k, proportionality constant, is:

0.70: for adolescent males  $\geq$  12 years old

0.55: for adolescent females  $\geq$  12 years old 0.55: for children (>=2 and <12 years old)

These baseline characteristics will be summarized using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) for continuous variables and using the numbers and percentages of subjects for categorical variables. The summary of baseline characteristics will be provided for the Safety Analysis Set.

A by-subject listing of other baseline characteristics will be provided by subject ID number in ascending order.

A separate by-subject data listing for prior HCV treatment and response will be provided for all subjects. The listing will display the prior HCV treatment experience for all subjects as well as the prior HCV regimen and treatment, the treatment duration, and the prior HCV treatment response for treatment experienced subjects.

#### 5.3. Swallowability Assessment for LDV/SOF Tablets

Swallowability Assessment (Able to swallow LDV/SOF FDC 90mg/400 mg or LDV/SOF FDC 22.5 mg/100 mg placebo tablet) will be summarized using the numbers and percentages of subjects in each swallowability category (ie, Able to Swallow, Unable to Swallow).

A by-subject listing of Swallowability of LDV/SOF FDC tablets will be provided by subject ID number in ascending order.

## 5.4. Medical History

General medical history (ie, conditions not specific to the disease being studied) data will be collected at screening and listed only. General medical history data will not be coded.

A by-subject listing of disease-specific medical history will be provided by subject ID number (in ascending order) and medical history of abnormalities (in chronological order).

## 6. EFFICACY ANALYSES

## 6.1. Primary Efficacy Endpoint

## 6.1.1. Definition of the Primary Efficacy Endpoint

The primary efficacy endpoint is SVR12 defined as HCV RNA < LLOQ (ie, < 50 IU/mL) 12 weeks after discontinuation of all study drugs in the FAS. The artus® HCV RG RT-PCR Kit by QIAGEN March 2015 are used to measure HCV RNA.

## 6.1.2. Primary Analysis of the Primary Efficacy Endpoint

The SVR12 rate in each of the HCV genotypes and overall will be calculated along with 2-sided 95% exact CI based on Clopper-Pearson method {20839}. No statistical hypothesis testing will be performed.

### 6.1.3. Subgroup Analysis of the Primary Efficacy Endpoint

Point estimates and 95% exact CIs of the SVR12 rates will be displayed for each subgroup outlined in Section 3.4.

A Forest plot will graphically present estimates and 95% CIs in SVR12 rates for each of the subgroups.

#### **6.2.** Secondary Efficacy Endpoints

## 6.2.1. Definition of Secondary Efficacy Endpoints

Secondary efficacy endpoints include the following:

- The proportion of subjects with HCV RNA < LLOQ at 4 and 24 weeks after discontinuation of treatment (SVR4 and SVR24)
- The proportion of subjects with HCV RNA < LLOQ while on treatment by study visit
- HCV RNA (log<sub>10</sub> IU/mL) and change from baseline in HCV RNA (log<sub>10</sub> IU/mL) through end of treatment (EOT)
- The proportion of subjects with virologic failure as the following:
- On-treatment virologic failure
  - HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ, while on treatment, confirmed with 2 consecutive values (note, second confirmation value can be posttreatment), or last available on-treatment measurement with no subsequent follow up values (ie, breakthrough)

- > 1 log<sub>10</sub>IU/mL increase in HCV RNA from nadir while on treatment, confirmed with 2 consecutive values (note, second confirmation value can be posttreatment), or last available on-treatment measurement with no subsequent follow up values (ie, rebound)
- o HCV RNA persistently ≥ LLOQ through 8 weeks of treatment (ie, nonresponse)

#### — Relapse

- HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA
   < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement</li>
- Characterization of HCV drug resistance substitutions at baseline, during, and after therapy with LDV/SOF

## 6.2.2. Analysis Methods for Secondary Efficacy Endpoints

For analyses of HCV RNA < LLOQ by visit while on treatment and during the posttreatment (SVR) follow-up period, subjects will be assigned a value at each visit based on the analysis visit windows specified in Section 3.7.2. Missing values will be imputed based on the categorical imputation rules described in Section 3.5.1. The 2-sided 95% exact confidence interval based on Clopper-Pearson method will be provided for the percentage of subjects with HCV RNA < LLOQ at each visit. The overall category for "HCV RNA < LLOQ" will be split into the following 2 subcategories: "< LLOQ TND" for subjects with target not detected and "< LLOQ detected" for subjects with < LLOQ detected in tabular displays.

Graphs for the percentage of subjects with HCV RNA < LLOQ over time during treatment will be displayed.

Summary statistics will be presented for absolute values and change from baseline in HCV RNA ( $log_{10}$  IU/mL) by visit through EOT. Imputation rules described in Section 3.5.1 will be used to assign HCV RNA values for missing values at a visit that are bracketed by "< LLOQ TND" and/or "< LLOQ detected". Otherwise, a missing = excluded analysis will be performed. Plots of the mean  $\pm$  SD and median (Q1, Q3) of absolute values and changes from baseline in HCV RNA through EOT will be presented.

For the SVR12 endpoint analysis, a summary table of the number and percentage of subjects with SVR12, virologic failure (VF), and Other will be created. All subjects who achieve SVR12 will be categorized as SVR12. Virologic failure will be descriptively summarized as "on-treatment virologic failure" and relapse (which will be broken down by study drug completed yes/no). Subjects who do not achieve SVR12 and do not meet criteria for VF will be categorized as Other. The denominator for relapse will be the number of subjects who had HCV RNA < LLOQ on their last observed on-treatment HCV RNA measurement; otherwise, the denominator will be the number of subjects in the FAS.

In addition, a summary table of the number and percentage of subjects with HCV RNA < LLOQ and >= LLOQ at the posttreatment follow-up visit (observed and imputed, with

reasons for imputed) will be provided for each posttreatment follow-up visit. 95% Clopper-Pearson exact CIs may be presented for the overall proportion of subjects with HCV RNA < LLOQ.

A concordance table between SVR12 and SVR24 will be provided. Subjects with both observed SVR12 and observed SVR24 data will be included for this analysis.

Drug resistant substitutions will be analyzed as part of the Virology Study Report.

## **Exploratory Endpoints of Interest**

## **6.3.1.** Definition of Exploratory Endpoints



## 6.3.2. Analysis Methods for Other Endpoints of Interest

PPD



## 6.4. Changes From Protocol-Specified Efficacy Analyses

There are no changes from protocol-specified efficacy analyses.

## 7. SAFETY ANALYSES

#### 7.1. Adverse Events and Deaths

#### 7.1.1. Adverse Event Dictionary

Clinical and laboratory adverse events (AEs) will be coded using the current version of MedDRA. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

## 7.1.2. Adverse Event Severity

Adverse events are graded by the investigator as Grade 1, 2, 3, or 4 according to toxicity criteria specified in the protocol. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings and the most severe will be considered (for sorting purpose only) in data presentation.

### 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE eCRF to the question of "Related to Study Treatment". Events for which the investigator did not record relationships to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing from that captured on the CRF.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if AEs met the definitions of SAE specified in the study protocol. Serious adverse events captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Drug Safety and Public Health Department before database finalization.

## 7.1.5. Treatment-Emergent Adverse Events

#### 7.1.5.1. Definition of Treatment Emergent

Treatment-emergent adverse events (TEAEs) are defined as one or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug.
- Any AEs leading to premature discontinuation of study drug.

#### 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent, as long as the AE

stop date is not prior to the first dose date of study drug. The event is considered treatment emergent if both of the following 2 criteria are met:

- The AE onset and end dates are the same as or after the month and year (or year) of the first dose date of study drug
- The AE onset date is the same as or before the month and year (or year) of the 30th day after the date of the last dose of study drug

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dose date of study drug, will be considered to be treatment emergent.

#### 7.1.6. Summaries of Adverse Events and Deaths

A brief high-level summary of TEAEs will be provided by the number and percentage of subjects who had the following: any AE; any AE of Grade 3 or above; any AE of Grade 2 or above; any treatment-related AE; any treatment-related AE of Grade 3 or above; any treatment-related AE of Grade 2 or above; any SAE; any treatment-related SAE; any AE that led to premature discontinuation of LDV/SOF (90mg/400mg) or LDV/SOF(22.5mg/100mg); any AE leading to interruption of LDV/SOF (90mg/400mg) or LDV/SOF(22.5mg/100mg). All deaths (including those that are treatment emergent and those that are not treatment emergent) observed during the study will also be summarized and included in this table.

Adverse event summaries will provide the number and percentage of subjects with TEAEs by SOC and PT, based on the Safety Analysis Set as follows:

- All AEs
- AEs of Grade 3 or above
- AEs of Grade 2 or above
- All treatment-related AEs
- Treatment-related AEs of Grade 3 or above
- Treatment-related AEs of Grade 2 or above
- All SAEs
- All treatment-related SAEs
- All AEs leading to premature discontinuation of LDV/SOF
- Deaths

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC and then by PT in order of descending incidence of the pooled treatment groups within each SOC. In summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual subject during the study.

In addition to the above summary tables, TEAEs will be summarized by PT only, in order of descending incidence for:

- AEs of Grade 3 or above
- All treatment-related AEs
- All SAEs
- AEs leading to premature discontinuation of LDV/SOF

In addition to the by-treatment summaries described above, data listings will be provided for the following:

- All AEs (with a variable indicating whether the event is treatment emergent)
- AEs of Grade 3 or above
- SAEs
- Deaths
- AEs leading to premature discontinuation of LDV/SOF

## 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the Safety Analysis Set and will include data collected up to the last dose of study drug plus 30 days for subjects who have permanently discontinued study drug or all available data at the time of the database snapshot for subjects those who were ongoing at the time of an interim analysis. The analysis will be based on values reported in conventional units. When values are below the limit of quantitation, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics. For example, if "< 0.2" was recorded, a value of 0.1 will be used for the purpose of calculating summary statistics; if "< 0.1" was recorded, a value of 0.09 will be used for the purpose of calculating summary statistics. Hemolyzed test results will not be included in the analysis, but they will be listed in by-subject laboratory listings.

A by-subject listing for laboratory test results will be provided by subject ID number and visit in chronological order for hematology, serum chemistry, and urinalysis separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or

higher on the Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities will be flagged in the data listings, as appropriate.

No inferential statistics will be generated.

#### 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) will be provided for ALT, aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase, hemoglobin, reticulocytes, white blood cell (WBC), neutrophils, lymphocytes, platelets, activated partial thromboplastin time (APTT), International Normalized Ratio of prothrombin time(INR), creatinine and CrCL (Schwartz formula) as follows:

- Baseline values
- Values at each postbaseline time visit
- Change from baseline at each postbaseline visit

A baseline laboratory value will be defined as the final assessment performed on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the visit value minus the baseline value. The mean, median, Q1, Q3, minimum, and maximum will be displayed to the reported number of digits; SD to the reported number of digits plus 1.

Median (Q1, Q3) of the observed values for ALT, AST, total bilirubin, alkaline phosphatase, creatinine, hemoglobin, reticulocytes, WBC, neutrophils, lymphocytes, and platelets will be plotted using a line plot by visit.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3 (Selection of Data in the Event of Multiple Records in a Window).

#### 7.2.2. APRI Calculation

AST to Platelet Ratio Index (APRI) is assessed at screening, week 12, Early Study Drug Discontinuation (ESDD) as applicable, and Post Treatment Week 4. APRI is derived by corresponding AST, platelet value with formula: [AST (U/L)/upper limit of normal (U/L)] × 100/platelets (10^9/L). Local lab National Cancer Institute, Egypt (NCI) ULN of AST is 46 U/L. Descriptive statistics and change from baseline will be provided.

## 7.2.3. Graded Laboratory Values

The Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities will be used for assigning toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. Some laboratory tests have criteria for both increased and decreased levels; analyses for each direction (ie, increased, decreased) will be presented separately.

## 7.2.3.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days for subjects who permanently discontinued study drug, or all available data in the database snapshot for subjects who were still on treatment at the time of an interim analysis. If the relevant baseline laboratory value is missing, then any abnormality of at least Grade 1 will be considered treatment emergent.

## 7.2.3.2. Summaries of Laboratory Abnormalities

Laboratory data that are categorical will be summarized using the number and percentage of subjects in the study with the given response at baseline and each scheduled postbaseline visit.

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by analyte and treatment group; subjects will be categorized according to the most severe postbaseline abnormality grade for a given analyte:

- Graded laboratory abnormalities
- Grade 3 or above laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with nonmissing postbaseline values up to 30 days after last dose for the laboratory parameter of interest.

A by-subject listing of treatment-emergent Grade 3 or above laboratory abnormalities will be provided by subject ID number and visit in chronological order. This listing will include all test results that were collected throughout the study for the analyte of interest, with all applicable severity grades or abnormal flags displayed.

## 7.3. Body Weight, Height, and Vital Signs

Vital signs (systolic and diastolic blood pressure [mmHg], pulse [beats/min]), body weight (kg), height (cm), and BMI(kg/m²) at each visit, and change from baseline at each visit will be summarized for the Safety Analysis Set using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum). The baseline value will be defined as the last available value collected on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.7.3 (Selection of Data in the Event of Multiple Records in a Window). No inferential statistics will be generated.

A by-subject listing of vital signs (systolic and diastolic blood pressure [mmHg], pulse [beats/min], respiration [breaths/min], and body temperature [°C]) will be provided by

subject ID number and visit in chronological order. In the same manner, a by-subject listing of body weight, height, and BMI will be provided separately.

#### 7.4. Prior and Concomitant Medications

Medications collected at screening and during the study will be coded using the current version of the World Health Organization (WHO) Drug dictionary.

#### 7.4.1. Prior Medications

Prior medications are defined as any medications taken before a subject took the first study drug.

#### 7.4.2. Concomitant Medications

Concomitant medications are defined as medications taken while a subject took study drug. Use of concomitant medications will be summarized by preferred name using the number and percentage of subjects for each treatment group. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered by generic name in descending overall frequency. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medications with a start date prior to or on the first dosing date of study drug and continued to be taken after the first dosing date, or started after the first dosing date but prior to or on the last dosing date of study drug will be considered concomitant medications. Medications started and stopped on the same day as the first dosing date or the last dosing date of study drug will also be considered concomitant. Medications with a stop date prior to the date of first dosing date of study drug or a start date after the last dosing date of study drug will be excluded from the concomitant medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the date of first study drug administration will be excluded from the concomitant medication summary. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) after the study drug stop date will be excluded from the concomitant medication summary. Medications with completely missing start and stop dates will be included in the concomitant medication summary, unless otherwise specified. Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

All prior and concomitant medications (other than per-protocol study drugs) will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order. Anatomical Therapeutic Chemical (ATC) drug class will not be listed.

#### 7.5. Other Safety Measures

A data listing for cirrhosis determination will be provided for all subjects at screening.

A data listing will be provided for subjects who become pregnant during the study.

No additional safety measures are specified in the protocol.

## 7.6. Changes From Protocol-Specified Safety Analyses

There are no deviations from the protocol-specified safety analyses.

## 8. PHARMACOKINETIC ANALYSES

No pharmacokinetics (PK) sample was collected. As such, no PK analysis is planned for this study.

| 9. | REFERENCES |
|---|---|
| 16978 | Koch GG, Carr GJ, Amara IA, Stokes ME, Uryniak TJ. Categorical Data<br>Analysis. Chapter 13 in Berry, D.A. (ed.). Statistical Methodology in the<br>Pharmaceutical Sciences. New York: Marcel Dekker, Inc., 1989:pp. 414-21. |
| 20503 | Chan IS, Zhang Z. Test-based exact confidence intervals for the difference of two binomial proportions. Biometrics 1999;55 (4):1202-9. |
| 20839 | Clopper CJ, Pearson ES. The Use of Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Biometrika 1934 Dec; 26 (4):pp. 404-13. |

## 10. SOFTWARE

SAS® Software Version 9.4. SAS Institute Inc., Cary, NC, USA.

## 11. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| - | | | |

## **APPENDICES**

12.

Appendix 1. Schedule of Assessments

## Appendix Table 1. Screening, On-Treatment Visits

| | Screening | Treatment | | | | | |
|---|---|---|---|---|---|---|---|
| | Day -28<br>to Day -1 | Baseline/<br>Day 1 <sup>a</sup> | Week 1<br>(±3 days) | Week 4<br>(±3 days) | Week 8<br>(±3 days) | Week 12<br>(±3 days) | ESDD |
| Consent /Assent | X | | | | | | |
| Demographics | X | | | | | | |
| Medical History | X | X | | | | | |
| Physical exam (PE) | X | | | | | | |
| Symptom directed PE | | X | X | X | X | X | X |
| Height and weight | X | X | | X | X | X | X |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X |
| Swallowability Assessment | X | | | | | | |
| AEs and Con-Meds | X | X | X | X | X | X | X |
| HBsAg, HBsAb, HBcAb, HIV antibody, HAV antibody, HCV antibody | X | | | | | | |
| HCV RNA | X | X | X | X | X | X | X |
| HCV genotype | X | | | | | | |
| HBV DNA ° | | X | | X | X | X | X |
| IL28B genotype | | X | | | | | |
| Urinalysis | X | | | | | | |
| Hematology and Blood Chemistry (including ALT) | X d | X | | X | X | X | X |

PPD


| | Screening | Treatment | | | | | |
|---|---|---|---|---|---|---|---|
| | Day -28<br>to Day -1 | Baseline/<br>Day 1 <sup>a</sup> | Week 1<br>(±3 days) | Week 4<br>(±3 days) | Week 8<br>(±3 days) | Week 12<br>(±3 days) | ESDD |
| Fibrotest | X | X | | | | X | X |
| FibroScan | X | | | | | | |
| APRI Calculation | X | | | | | X | X |
| Coagulation | X | X | | | | X | X |
| Pregnancy test <sup>e</sup> | X | X | | X | X | X | X |
| Pregnancy prevention counseling <sup>f</sup> | | X | | | | X | X |
| Dispense drug | | X | | X | X | | |
| Review subject dosing diary | | X | X | X | X | X | |
| Review of Study Drug Adherence and Drug<br>Accountability | | | X | X | X | X | X |

a Baseline/Day 1 assessments must be performed prior to dosing.


b Vital signs include resting blood pressure, pulse, respiratory rate, and temperature. SAE and study procedure related AEs are to be collected form informed consent. Other AEs are to be collected from Baseline/Day1.

c HBV DNA testing done only when subjects are HBcAb positive at Screening

For females of childbearing potential only: serum β-hCG at Screening, urine test thereafter. If urine is positive, confirm immediately with serum β-hCG

f If applicable

## Appendix Table 2. Post-Treatment Study Visits

| | 4 Weeks Post-Treatment<br>(±5 days) | 12 Weeks Post-Treatment <sup>a</sup><br>(±5 days) | 24 Weeks Post-Treatment<br>(±5 days) |
|---|---|---|---|
| Clinical Assessments | | | |
| Symptom-directed PE | X | | |
| Height and Weight | X | X | X |
| Vital Signs | X | | |
| AEs | X | $X^a$ | Xa |
| Concomitant Medications | X | | |
| Fibrosis assessment <sup>b</sup> | | X | X |
| Pregnancy prevention counseling <sup>c</sup> | X | | |
| Laboratory Assessments | | | |
| Hematology and Blood Chemistry | X | | X |
| APRI Calculation | X | | |
| HCV RNA | X | X | X |
| HBV DNA <sup>d</sup> | X | X | X |
| PPD | | | |
| Urine Pregnancy Test <sup>f</sup> | X | | |

a All SAEs, including deaths, regardless of cause or relationship, must be reported after patient signs the informed consent through the end of the study

f Females of childbearing potential


b Fibroscan and Fibrotest

c If applicable

d HBV DNA testing done only when subjects are HBcAb positive at Screening